CLINICAL TRIAL: NCT04002700
Title: Stroke Risk Among Users of Typical vs. Atypical Antipsychotics Stratified by Broad Age Group, a Post-authorization Safety Study
Brief Title: A Study to Assess Stroke Risk Among Users of Typical Versus Atypical Antipsychotics Stratified by Broad Age Group
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108624; PCSESP001292 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Haloperidol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (9):
- Target Cohort 1: Participants will be analyzed for stroke-risk who are new users of typical antipsychotics aged 18 to 64 years without a recent dementia diagnosis.
  Interventions: Drug: Typical Antipsychotics
- Target Cohort 2: Participants will be analyzed for stroke-risk who are new users of haloperidol aged 18 to 64 years without a recent dementia diagnosis.
  Interventions: Drug: Haloperidol
- Target Cohort 3: Participants will be analyzed for stroke-risk who are new users of typical antipsychotics aged greater than or equal to (>=) 65 years.
  Interventions: Drug: Typical Antipsychotics
- Target Cohort 4: Participants will be analyzed for stroke-risk who are new users of haloperidol aged >= 65 year.
  Interventions: Drug: Haloperidol
- Target Cohort 5: Participants will be analyzed for stroke-risk who are new users of typical antipsychotics aged 18 to 64 years.
  Interventions: Drug: Typical Antipsychotics
- Target Cohort 6: Participants will be analyzed for stroke-risk who are new users of haloperidol aged 18 to 64 years.
  Interventions: Drug: Haloperidol
- Comparator Cohort 7: Participants will be analyzed for stroke-risk who are new users of atypical antipsychotics aged 18-64 years without a recent dementia diagnosis.
  Interventions: Drug: Atypical Antipsychotics
- Comparator Cohort 8: Participants will be analyzed for stroke-risk who are new users of atypical antipsychotics aged >= 65 years.
  Interventions: Drug: Atypical Antipsychotics
- Comparator Cohort 9: Participants will be analyzed for stroke-risk who are new users of atypical antipsychotics aged 18-64 years.
  Interventions: Drug: Atypical Antipsychotics

INTERVENTIONS:
Drug: Haloperidol — Stroke rates among participants from 01 January, 2002 through 31 December 2017 will be estimated among new users of haloperidol. No drug will be administered as part of this study.
  Groups: Target Cohort 2; Target Cohort 4; Target Cohort 6
Drug: Typical Antipsychotics — Stroke rates among participants from 01 January, 2002 through 31 December 2017 will be estimated among new users of typical antipsychotics which includes Haloperidol, Loxapine, Thioridazine, Molindone, Thiothixene, Fluphenazine, Trifluoperazine, Perphenazine, Chlorpromazine. No drug will be administered as part of this study.
  Groups: Target Cohort 1; Target Cohort 3; Target Cohort 5
Drug: Atypical Antipsychotics — Stroke rates among participants from 01 January, 2002 through 31 December 2017 will be estimated among new users of atypical antipsychotics which includes Aripriprazole, Asenapine, Brexpiprazole, Cariprazine, Clozapine, Iloperidone, Lurasidone, Paliperidone, Ziprasidone, Risperidone, Quetiapine, Olanzapine. No drug will be administered as part of this study.
  Groups: Comparator Cohort 7; Comparator Cohort 8; Comparator Cohort 9

SUMMARY:
The purpose of this study is to extend the recent Food and Drug Administration (FDA) Sentinel tabulations regarding stroke risk among new users of typical and atypical antipsychotics to participants who were aged 18-64 years and did not have dementia to participants aged 65 years and older regardless of dementia status.

ELIGIBILITY:
Inclusion Criteria:

For entry event of an initial drug exposure:

* First exposure to the particular drug(s) in the past 183 days (index date)
* Had at least 183 days of continuous observation time prior to index
* Exactly 0 condition occurrences of 'Cancer' any time in the 183 days before or on the index date
* Exactly 0 condition occurrences of 'Stroke' any time in the 183 days before or on the index date
* Exactly 0 exposures to any other typical or atypical antipsychotics any time in the 183 days before or on the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is the participants in (any of) the target or comparator cohorts. Each target and comparator cohort will be drawn from the appropriate database: IBM MarketScan Commercial Database (CCAE) if the participants are aged 18-64 years and IBM MarketScan Medicare Supplemental Database (MDCR) if participants are aged greater than or equal to (>=) 65 years.
Sampling Method: Probability Sample
Enrollment: 1234412 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Stroke as a Principal Inpatient Diagnosis | Up to 16 years (from 01-January-2002 through 31-December-2017)
  Number of participants with stroke in each target cohort versus comparator cohort (aged 65 years and older) per person years at risk will be reported. It is defined defined by the presence of the relevant ICD codes (ICD-9 or ICD-10 according to date) in the inpatient setting as the primary diagnoses.

SECONDARY OUTCOMES:
Number of Participants at Stroke Risk when Compared Among New Users of Typical Antipsychotics/Haloperidol versus Atypical Antipsychotics | Up to 16 years (from 01-January-2002 through 31-December-2017)
  The number of participants with the risk of stroke among participants exposed to typical antipsychotics versus atypical antipsychotics will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Janssen Investigative Site, Titusville, New Jersey, United States